CLINICAL TRIAL: NCT04346563
Title: Effect of Kinesio Taping on Upper Extremity Performance in Individuals With Rounded Shoulders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTMahidolU1
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Shoulder Pain
Keywords: Kinesio tape, Functional correction, Rounded shoulder
MeSH Terms: conditions — Shoulder Pain | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: RCT among two groups,
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocated participants, they do not know which group they would be in. Assessor do not know which group of participant that would perform.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio tape, functional correction applying (Experimental): The experimental group, trained by Certified Kinesio tape researcher will attache the kinesio tape. Attaching the kinesio tape by using functional correction techniques, apply tape from the front of the acromion process to the spinous process T10 on both sides, providing 50% of the tape's tension (Kase, 2003, Han JT et al) to create a scapular retraction.
  Interventions: Other: Kinesio tape, functional correction technique; Other: Elastic band strengthening shoulder exercise
- Placebo Kinesio taping apply (Placebo Comparator): Apply kinesio tape without tension.
  Interventions: Other: Elastic band strengthening shoulder exercise

INTERVENTIONS:
Other: Kinesio tape, functional correction technique — According to Kinesio Taping, functional correction technique could use for correcting shoulder, scapular alignment and decrease pain.
  Arms: Kinesio tape, functional correction applying
Other: Elastic band strengthening shoulder exercise — The exercise in which both groups will receive Introduction of exercise with rubber bands (Elastic band) It is a home exercise (Home base exercise program) for patients to do with appropriate resistance. Which can be done at least 10 times and not more than 20 times continuously,will be asked to do all 3 positions.
  1) Shoulder external rotation in shoulder abduction 90 degrees 2) Shoulder horizontal abduction in shoulder abduction 90 degrees 3) Seated bend row, which will be done 15 times, each hold for 10 seconds, do 3 sets, each set rest 2 minutes, 2 times a day ( Morning-evening) consecutively for 1 week

SUMMARY:
The objective of this research is to study the effect of kinesio tapes with functional correction technique in combination with exercise management to increase strength and decrease pain, in people with rounded shoulders. The study would be evaluated with the EvaltechTM machine, (functional capacity assessment).

DETAILED DESCRIPTION:
Participants

* Age 25-50 years, male and female
* People who have a shoulder condition. (By measuring in the supine position, distance from the posterior aspect of acromion to the bed> 1 inch on both sides)
* People with moderate to severe neck and shoulder pain (VAS> 3)
* People who have to use their arms for work Overall more than 3 hours per day

For attaching the tape, the researcher will prepare a replacement shirt in case the For the convenience of tape, the experimental group, trained by Certified Kinesio tape, attached the kinesio tape. Attaching the tape By using functional correction techniques, apply from the front of the acromion process to the spinous process T10 on both sides.

Measurements

1. The pressure of (average of peak force) of both arms (pounds)
2. The pulling force (average of peak force) of both arms (pounds)
3. Time of overhead endurance test (TMT) (seconds)
4. Visual analog scale (VAS)
5. The distance from the posterior aspect of acromion to the bed (inches)

process of measuring the evaluation 3 times

1. st after physical therapy treatment Before attaching the kinase tape
2. nd evaluation period was 48 hours apart before the next treatment.
3. rd evaluation period is 1 week apart.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-50 years, male and female
* People who have a shoulder condition. (By measuring in the supine position, distance from the posterior aspect of acromion to the bed> 1 inch on both sides)
* People with moderate to severe neck and shoulder pain (VAS> 3)
* People who have to use their arms for work Overall more than 3 hours per day

Exclusion Criteria:

* People with neck pain, fracture in the arm, and numbness
* People who have pain and have limited shoulder movement of the shoulder joint
* People who have had a history of spine / shoulder surgery
* People with a history of allergies to cloth tapes
* People who have rheumatoid arthritis that affects inflammation of the joints such as rheumatoid etc.
* People receiving medication that affects their participation in the study
* People with neurological symptoms
* People with cognitive disabilities

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The pushing force (average of peak force) of both arms (pounds) | 2 minutes
  Maximum strength of pushing, measures by Evaltech machine
The pulling force (average of peak force) of both arms (pounds) | 2 minutes
  Maximum strength of pulling, measures by Evaltech machine
Time measurement tolerance (TMT) (seconds) | 4 minutes
  Time tolerance of overhead reaching, measures by Evaltech machine

SECONDARY OUTCOMES:
Visual analog pain scale (VAS) | 1 minute
  0-10 centimeters visual analog scale, higher score means higher pain and worse outcome
The distance from the posterior aspect of acromion to the bed (inches) | 2 minutes
  Measure in lying position by measurement tape

CONTACTS AND LOCATIONS:
Overall Officials: Prasert Sakulsriprasert, PhD, Principal Investigator — Lecturer
Locations (1):
- Mahidol University, Salaya, Nakhonpathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han JT, Lee JH, Yoon CH. The mechanical effect of kinesiology tape on rounded shoulder posture in seated male workers: a single-blinded randomized controlled pilot study. Physiother Theory Pract. 2015 Feb;31(2):120-5. doi: 10.3109/09593985.2014.960054. Epub 2014 Sep 29. PMID 25264014
- [Background] El-Abd AM, Ibrahim AR, El-Hafez HM. Efficacy of kinesiology tape versus postural correction exercises on neck disability and axioscapular muscles fatigue in mechanical neck dysfunction: A randomized blinded clinical trial. J Bodyw Mov Ther. 2017 Apr;21(2):314-321. doi: 10.1016/j.jbmt.2016.07.008. Epub 2016 Jul 26. PMID 28532874
- [Background] Ay S, Konak HE, Evcik D, Kibar S. The effectiveness of Kinesio Taping on pain and disability in cervical myofascial pain syndrome. Rev Bras Reumatol Engl Ed. 2017 Mar-Apr;57(2):93-99. doi: 10.1016/j.rbre.2016.03.012. Epub 2016 May 10. English, Portuguese. PMID 28343625
- [Background] Kim MK, Lee JC, Yoo KT. The effects of shoulder stabilization exercises and pectoralis minor stretching on balance and maximal shoulder muscle strength of healthy young adults with round shoulder posture. J Phys Ther Sci. 2018 Mar;30(3):373-380. doi: 10.1589/jpts.30.373. Epub 2018 Mar 2. PMID 29581654
- [Background] Kim TW, An DI, Lee HY, Jeong HY, Kim DH, Sung YH. Effects of elastic band exercise on subjects with rounded shoulder posture and forward head posture. J Phys Ther Sci. 2016 Jun;28(6):1733-7. doi: 10.1589/jpts.28.1733. Epub 2016 Jun 28. PMID 27390405
- [Background] Peppers D, Figoni SF, Carroll BW, Chen MM, Song S, Mathiyakom W. Influence of Functional Capacity Evaluation on Physician's Assessment of Physical Capacity of Veterans With Chronic Pain: A Retrospective Analysis. PM R. 2017 Jul;9(7):652-659. doi: 10.1016/j.pmrj.2016.10.011. Epub 2016 Oct 22. PMID 27780768